CLINICAL TRIAL: NCT04876807
Title: A Phase 1, Single-center, Open-label, Fixed-sequence, 4-period, 3-part Study in Healthy Adult Subjects to Evaluate the Effect of an Acidic Formulation of Acalabrutinib (ACP-196), Acidic Beverage, or Grapefruit Juice on the Pharmacokinetics of Acalabrutinib Alone and Coadministered With Omeprazole
Brief Title: A Study to Evaluate the Effect of an Acidic Formulation of Acalabrutinib (ACP-196), Acidic Beverage, or Grapefruit Juice on the Pharmacokinetics (PK) of ACP-196 Alone and Coadministered With Omeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HV-112
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: Acalabrutinib; ACP-196; Healthy volunteers; Pharmacokinetics; PK; Acidic Formulation; Acidic Beverage; Grapefruit Juice; Omeprazole; Fixed-sequence
MeSH Terms: interventions — acalabrutinib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Acidic formulation) (Experimental): In Part 1 of the study, the participants will receive Dose 1 of ACP-196 (reference or acidic formulation as applicable) with 240 mL water in 4 treatment schedules on Day 1, Day 3, Day 8 (with omeprazole), and Day 10 (with omeprazole).
  Interventions: Drug: ACP-196; Drug: Omeprazole
- Part 2 (Orange drink) (Experimental): In Part 2 of the study, the participants will receive Dose 1 of ACP-196 (reference formulation) with 240 mL water or acidic beverage as applicable in 4 treatment schedules on Day 1, Day 3, Day 8 (with omeprazole), and Day 10 (with omeprazole).
  Interventions: Drug: ACP-196; Drug: Omeprazole
- Part 3 (Grapefruit juice) (Experimental): In Part 3 of the study, the participants will receive Dose 1 of ACP-196 (reference formulation) with 240 mL water or grapefruit as applicable in 4 treatment schedules on Day 1, Day 3, Day 8 (with omeprazole), and Day 10 (with omeprazole).
  Interventions: Drug: ACP-196; Drug: Omeprazole

INTERVENTIONS:
Drug: ACP-196 — In Parts 1, 2, and 3, participants will receive oral Dose 1 of ACP-196 (reference or acidic formulation as applicable) on Day 1, Day 3, Day 8, and Day 10.
  Other Names: Acalabrutinib
Drug: Omeprazole — Participants will receive omeprazole in all parts as: on Day 8 and Day 10 with water in Part 1; on Day 8 with water and on Day 10 with acidic beverage in Part 2; on Day 8 with water and on Day 10 with grapefruit juice in Part 3.

SUMMARY:
This study will evaluate the effect of an acidic formulation of Acalabrutinib (ACP-196), acidic beverage, or grapefruit Juice on the PK of ACP-196 alone and coadministered with omeprazole.

DETAILED DESCRIPTION:
This is a 3-part study. Each part of the study will compare the effect of an acidic formulation of ACP-196, acidic beverage (orange drink), or grapefruit juice on the PK profile of ACP-196 alone and when coadministered with omeprazole. Participants will be enrolled into Part 1 of the study first and then subsequent participants will be randomized in a 1:1 ratio to either Part 2 or Part 3 of the study. Participants will be screened within 28 days before the dose. Participants will be contacted approximately 14 days after the last dose of study drug administration to determine if any adverse event has occurred since the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker who has not used nicotine-containing products for ≥ 3 months before the first dose.
* Body mass index (BMI) >= 18.0 and =< 32.0 kg/m^2 at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms, as deemed by the principal investigator (PI). Liver function tests must be =< the upper limit of normal range (ULN) at screening for inclusion.
* Men and women of reproductive potential to follow protocol defined contraception methods.
* Women must have negative serum pregnancy test results.
* Willing and able to take the study drug with 240 mL of orange drink (Part 2) or grapefruit juice (Part 3).

Exclusion Criteria:

* Participant is mentally or legally incapacitated, or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* Participant with known fruit allergies.
* History or presence of clinically significant medical or psychiatric condition or disease (eg, cardiovascular, respiratory, hepatic, gastrointestinal, renal, genitourinary, endocrine, neuromuscular, rheumatologic, oncologic, cutaneous or other disorders), in the opinion of the PI.
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* Presence of any clinically significant, ongoing systemic bacterial, fungal or viral infections in the opinion of the PI.
* History or presence of alcoholism or drug abuse within the past 2 years before screening.
* History of bleeding diathesis (eg, hemophilia, von Willebrand disease).
* Any clinically significant condition that may affect acalabrutinib absorption in the opinion of the PI, including gastric restrictions and bariatric surgery (eg, gastric bypass).
* History or presence of clinically significant thyroid disease, in the opinion of the PI.
* Women who are pregnant or breastfeeding.
* Positive urine drug or alcohol results at screening or check-in.
* Positive urine cotinine at screening.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Seated blood pressure is < 90/40 mm Hg or > 140/90 mm Hg at screening.
* Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
* Have been on a diet incompatible with the on study diet, in the opinion of the PI, within the 28 days before the first dose of study drug, and throughout the study.
* Unable to refrain from or anticipates the use of protocol defined medicines:
* Donation of blood or significant blood loss within 56 days before the first dose of study drug.
* Plasma donation within 7 days before the first dose of study drug.
* Prior exposure to acalabrutinib (ACP-196).
* History or presence of clinically significant hypersensitivity or idiosyncratic reaction to acalabrutinib, omeprazole, related compounds (eg, substituted benzimidazoles, other azole compounds), or any inactive ingredients.
* History or presence of liver disease and Clostridium difficile-associated diarrhea.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-last) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Maximum Observed Plasma Concentration (Cmax) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10

SECONDARY OUTCOMES:
Percent of AUC0inf Extrapolated (AUC%extrap) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours (AUC0-6h) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours (AUC0-12h) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Time to Reach Maximum Observed Plasma Concentration (Tmax) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Apparent Terminal Elimination Rate Constant (λz) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Apparent Terminal Elimination Half-life (T1/2) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Apparent Total Plasma Clearance (CL/F) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Apparent Total Volume of Distribution (Vz/F) of ACP-196 in Parts 1, 2, and 3 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 14, and 24 hours on Days 1, 3, 8, and 10
Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC0-24h) of Omeprazole in Parts 1, 2, and 3 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours on Days 8 and 10
Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-last) of Omeprazole in Parts 1, 2, and 3 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours on Days 8 and 10
Maximum Observed Plasma Concentration (Cmax) of Omeprazole in Parts 1, 2, and 3 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours on Days 8 and 10
Time of the Maximum Measured Plasma Concentration (Tmax) of Omeprazole in Parts 1, 2, and 3 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours on Days 8 and 10
Apparent Total Plasma Clearance (CL/F) of Omeprazole in Parts 1, 2, and 3 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours on Days 8 and 10
Apparent Total Volume of Distribution (Vz/F) of Omeprazole in Parts 1, 2, and 3 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, and 24 hours on Days 8 and 10
Number of Participants With Treatment emergent Adverse Events (TEAEs) and Treatment emergent Serious Adverse Events (TESAEs) in Parts 1, 2, and 3 | From Day 1 through 14 days after the last dose (approximately 2 months)
Number of Participants With Abnormal Vital Signs and Physical Examinations Reported as TEAEs in Parts 1, 2, and 3 | From Day 1 through 24 hours post last dose on Day 10 (approximately 2 months)
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in Parts 1, 2, and 3 | From Day 1 through 24 hours post last dose on Day 10 (approximately 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Priti Patel, MD, Study Director — Acerta Pharma BV
Locations (1):
- Laura Sterling, MD, MPH, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home